CLINICAL TRIAL: NCT05426720
Title: Risk Factors and Biomarkers for Post-tuberculosis Lung Damage in a Chinese Cohort: Protocol for a Prospective Observational Study
Brief Title: Risk Factors and Biomarkers for Post-tuberculosis Lung Damage
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Geriatric Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2022296
Record Dates: First submitted 2022-06-08; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Pulmonary TB
Keywords: post-tuberculosis lung damage; cigarette smoking
MeSH Terms: conditions — Tuberculosis, Pulmonary; Cigarette Smoking

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum cytokines including IL-6, IL-8, MMP and etc will be detected at baseline prior to TB treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with pulmonary tuberculosis: male patients aged 25-60 with active pulmonary tuberculosis
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention; This study is a observational study. All patients received routine anti-tuberculosis regimen. Researchers will observe the clinical manifestation, pulmonary function and pulmonary CT manifestation within a few years after the cure of tuberculosis.

SUMMARY:
This prospective study aims to determine the incidence of Post-tuberculosis lung damage (PTLD), examine trends in the changes in lung function, and investigate the impact of smoking and other factors on respiratory symptoms, lung function, and chest CT findings, which will aid in the development of prognostic and therapeutic strategies for PTLD.

DETAILED DESCRIPTION:
Introduction: Post-tuberculosis lung damage (PTLD) refers to residual pulmonary impairment following the completion of tuberculosis (TB) treatment, characterized by persistent respiratory symptoms and abnormal pulmonary function. The risk factors and biomarkers for PTLD have been scarcely investigated. Additionally, it remains unclear whether and to what extent cigarette smoking affects PTLD in patients with TB.

Methods and analysis: This prospective observational study will enroll 400 adult male ever-smoker or never-smoker patients aged 25-60 years, with newly confirmed active TB between 2022 and 2024 from the Department of Respiratory and Critical Care Medicine at Peking University Third Hospital and the Tuberculosis Department at Beijing Geriatric Hospital. Baseline data (age, smoking history, and smoking pack-years), clinical symptoms, lung functions, and chest CT (computed tomography) findings will be prospectively collected. Respiratory questionnaires, lung function measurements, and chest CT examinations will be completed during follow-up visits at 6 months after the initiation of TB treatment, immediately at the completion of TB treatment, and at 1 year, 2 years, and 3 years after the completion of TB treatment. Peripheral blood samples will be obtained at baseline to measure inflammatory mediators and cytokines in serum. The collected data will be analyzed to determine the incidence of and factors/biomarkers for PTLD after TB treatment.

ELIGIBILITY:
Inclusion Criteria:

Male patients aged 25-60 years newly diagnosed with active pulmonary TB.

Exclusion Criteria:

1. patients with positive sputum smear or TB culture results;
2. human immunodeficiency virus-positive patients;
3. patients infected with multidrug-resistant TB;
4. patients with malignant neoplasms (e.g., lung cancer) or severe cardiovascular and cerebrovascular diseases;
5. non-compliant patients who were unable to complete the lung function tests;
6. patients without lung parenchymal destruction (such as tuberculous pleurisy). -

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — self-representation of gender identity
Study Population: This prospective observational study will enroll male patients who were newly diagnosed with active TB from the Department of Respiratory and Critical Care Medicine at Peking University Third Hospital and the Tuberculosis Department at Beijing Geriatric Hospital between January 2022 and December 2024.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
lung function | half a year, 1 year, 2 year, and 3-year follow-up
  Forced expiratory volume (FEV1, l/min), and forced vital capacity (FVC,l/min) are the important parameters in lung function. FEV1/FVC, diffusing capacity for carbon monoxide (DLCO), and other indicators, will also be observed during follow-up.

SECONDARY OUTCOMES:
Absorption of TB lesions on lung CT scans after TB treatment | half a year, 1 year, 2 year, and 3year follow-up
  Chest CT images will be interpreted by a respiratory physician and a radiologist. Parenchymal and airway lesions detected on CT scans will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Sun, MD, Study Director — Respiratory and Critical Care Department, Peking University Third Hospital
Locations (2):
- China (2):
  - Peking University Third Hospital, Beijing
  - Beijing Geriatric Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided
We will discuss if the data of individuals after the completion of the study.

DOCUMENTS (1):
  • Study Protocol (2022-06-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT05426720/Prot_000.pdf